CLINICAL TRIAL: NCT00836095
Title: A Randomized Controlled Trial Comparing the ProSeal Laryngeal Mask Airway With the Laryngeal Mask Airway Supreme in Mechanically Ventilated Patients
Brief Title: Comparison of ProSeal Laryngeal Mask Airway to Laryngeal Mask Airway Supreme
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Sonia Vaida, M.D, Vice Chair for Research, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB 29920
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-03

CONDITIONS: Adverse Effect of Unspecified General Anesthetics
Keywords: laryngeal mask, proseal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supreme LMA (Other): Supreme Laryngeal mask airway is a new, single use laryngeal mask airway variant.
  The choice of the airway device will be randomized by opening a sealed envelope immediately before induction. The airway device will be blindly inserted by an experienced attending anesthesiologist.
  Interventions: Device: Supreme Laryngeal mask airway
- Proseal LMA (Active Comparator): Proseal is a multiple use, variant of the laryngeal mask airway.
  The choice of the airway device will be randomized by opening a sealed envelope immediately before induction. The airway device will be blindly inserted by an experienced attending anesthesiologist.
  Interventions: Device: Proseal laryngeal mask airway

INTERVENTIONS:
Device: Supreme Laryngeal mask airway — Supreme Laryngeal mask airway is a new, single use laryngeal mask airway variant
  Arms: Supreme LMA
Device: Proseal laryngeal mask airway — Proseal is a multiple use, variant of the laryngeal mask airway
  Arms: Proseal LMA

SUMMARY:
Laryngeal mask airway is a widely used device in routine anesthesia for airway management during surgery. It consists of a tube with an inflatable cuff that is inserted into the mouth after induction of general anesthesia. The Proseal Laryngeal mask airway and the Laryngeal mask airway Supreme are two variants of the Laryngeal mask airway. The laryngeal mask airway Supreme is a newer version of the laryngeal mask airway.

The research is being done to compare two variants of the laryngeal mask airway: the Proseal laryngeal mask airway and the Laryngeal mask airway Supreme. This study will determine if the newer model, the Laryngeal mask airway Supreme, is easier to insert and is better positioned than the older model, the Proseal laryngeal mask airway. Both models are approved for use by the FDA, and are routinely used to assure the airway during general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 75 years
* ASA I and II
* Mallampatti class: I and II
* Thyromental distance > than 6.5 cm
* Interincisor distance > than 3 cm
* BMI < 35 Kg/m2
* Patients scheduled to undergo anesthesia with an LMA for minor extraperitoneal surgical procedures in supine position

Exclusion Criteria:

* Weight < 50 kg
* BMI > 35 Kg/m2
* Pregnant patients
* Known or expected difficult airway
* Patients with active, untreated and unresolved gastroesophageal reflux
* Esophageal pathology, pulmonary pathology
* Laparoscopic procedures
* ENT procedures, gastrointestinal procedures, intraperitoneal surgical procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-01; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonia J Vaida, MD, Principal Investigator — Penn State
Locations (1):
- PennState Hershey Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Supreme LMA: Supreme Laryngeal mask airway: The Supreme Laryngeal mask airway is a new, single use laryngeal mask airway variant.
  The choice of the airway device will be randomized by opening a sealed envelope immediately before induction. The airway device will be blindly inserted by an experienced attending anesthesiologist.
- Proseal LMA: Proseal laryngeal mask airway: The Proseal is a multiple use, variant of the laryngeal mask airway.
  The choice of the airway device will be randomized by opening a sealed envelope immediately before induction. The airway device will be blindly inserted by an experienced attending anesthesiologist.
Period: Overall Study
Arm/Group | Supreme LMA | Proseal LMA
Started | 22 | 30
Completed | 22 | 27
Not Completed | 0 | 3
Not completed — Physician Decision | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Supreme LMA: The choice of the airway device will be randomized by opening a sealed envelope immediately before induction. The airway device will be blindly inserted by an experienced attending anesthesiologist.
  Supreme Laryngeal mask airway: Supreme Laryngeal mask airway is a new, single use laryngeal mask airway variant.
- Proseal LMA: The choice of the airway device will be randomized by opening a sealed envelope immediately before induction. The airway device will be blindly inserted by an experienced attending anesthesiologist.
  Proseal laryngeal mask airway: Proseal is a multiple use, variant of the laryngeal mask airway
- Total: Total of all reporting groups
Arm/Group | Supreme LMA | Proseal LMA | Total
Number analyzed (Participants) | 22 | 30 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (14) | 41 (14) | 45 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 32
  Male | 8 | 12 | 20

OUTCOME MEASURES:

1. Primary Outcome: Insertion Time
Description: The insertion time will be the measured time that it takes the anesthesiologist to insert the airway and verify ventilation of the patient's airway. Data reported will be time in seconds ± the standard deviation.
Time Frame: During intubation of the patient
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Supreme LMA: Supreme Laryngeal mask airway: The Supreme Laryngeal mask airway is a new, single use laryngeal mask airway variant
  The choice of the airway device will be randomized by opening a sealed envelope immediately before induction. The airway device will be blindly inserted by an experienced attending anesthesiologist.
- Proseal LMA: Proseal laryngeal mask airway: The Proseal is a multiple use, variant of the laryngeal mask airway
  The choice of the airway device will be randomized by opening a sealed envelope immediately before induction. The airway device will be blindly inserted by an experienced attending anesthesiologist.
Arm/Group | Supreme LMA | Proseal LMA
Number analyzed (Participants) | 22 | 27
seconds | 26 (10) | 18 (6)

2. Secondary Outcome: Insertion Success Rate
Description: Insertion success rate will be reported as the number of patients for whom the airway device was successfully inserted and ventilation was verified.
Time Frame: During intubation of the patient
Measure: Number; unit: Number of successful airway insertions
Arm/Group | Supreme LMA | Proseal LMA
Number analyzed (Participants) | 22 | 27
Number of successful airway insertions | 22 | 27

ADVERSE EVENTS:
Groups:
- Supreme LMA: Supreme Laryngeal mask airway is a new, single use laryngeal mask airway variant.
  The choice of the airway device will be randomized by opening a sealed envelope immediately before induction. Both airway devices will be blindly inserted by an experienced attending anesthesiologist.
  Supreme Laryngeal mask airway: Supreme Laryngeal mask airway is a new, single use laryngeal mask airway variant
- Proseal LMA: Proseal is a multiple use, variant of the laryngeal mask airway.
  The choice of the airway device will be randomized by opening a sealed envelope immediately before induction. Both airway devices will be blindly inserted by an experienced attending anesthesiologist.
  Proseal laryngeal mask airway: Proseal is a multiple use, variant of the laryngeal mask airway
Arm/Group | Supreme LMA | Proseal LMA
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/30
Other Adverse Events (participants affected / at risk) | 0/22 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No